CLINICAL TRIAL: NCT03009292
Title: Pharmacokinetic Study of E7080/Lenvatinib in Chinese Subjects With Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-C086-108
Record Dates: First submitted 2016-12-31; First posted 2017-01-04 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-03

CONDITIONS: Solid Tumor
Keywords: solid tumor; Lenvatinib; pharmacokinetics
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 24 mg lenvatinib (Experimental): Participants will receive once daily oral dosing of lenvatinib 24 milligrams (mg)
  Interventions: Drug: lenvatinib

INTERVENTIONS:
Drug: lenvatinib — once daily continuous dosing

SUMMARY:
Study E7080-C086-108 is an open-label, single- and multiple-dose pharmacokinetic (PK) study of lenvatinib (administered orally, once a day [QD]) in Chinese participants with solid tumor. A total of 12 participants will be enrolled to evaluate the PK of 24 milligrams (mg) QD dosing of lenvatinib.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a histological and/or cytological diagnosis of solid tumor
* Participants with solid tumor that is resistant to standard anti-tumor therapies, or for which no appropriate treatment is available
* Participants whose toxicity of previous treatment has recovered to Grade 1 or lower (except for alopecia)
* Participants who have completed previous anti-tumor therapy (such as surgery, radiotherapy) at least 4 weeks before treatment
* Participants who are 18 years or older at the time of obtaining informed consent
* Participants with an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 1
* Participants who meet all of the following items:

  * Hemoglobin ≥9.0 grams per deciliter (g/dL)
  * Neutrophil count ≥1.5×10^3/microliters (µL)
  * Platelet count ≥10×10^4/µL
  * Total bilirubin ≤1.8 milligrams (mg)/dL
  * Aspartate aminotransferase (AST) ≤100 International Units per liter (IU/L)
  * Alanine aminotransferase (ALT) ≤100 IU/L
  * Serum creatinine ≤1.5 mg/dL or creatinine clearance ≥50 milliliters per minute (mL/min). Creatinine clearance will be calculated based on Cockcroft-Gault method using the following formula: Male: (140-age) × weight ÷ (serum creatinine × 72); Female: 0.85 × (140-age) × weight ÷ (serum creatinine × 72).
* Participants expected to survive for 12 weeks or longer
* Males and females of childbearing potential must agree to use appropriate contraception from the giving of consent to 30 days after study drug administration. Female participants of childbearing potential must test negative for pregnancy at screening
* Participants who voluntarily agree to participate in this study in writing

Exclusion Criteria:

* Participants with brain metastasis accompanied by clinical symptoms or requiring treatment
* Participants with the following complications or medical history

  1. Systemic severe infections requiring medical treatment
  2. The following cardiovascular diseases

     1. Ischemic cardiac disease or arrhythmia requiring medical treatment
     2. Angina pectoris or myocardial infarction within 24 weeks before enrollment
     3. Corrected QT interval (QTc) greater than 480 milliseconds (msec) (Fridericia's method)
  3. Hemoptysis (fresh blood) ≥ 1/2 teaspoon (2.5 mL) or clinically significant hemorrhagic or thrombotic events within 4 weeks before enrollment
  4. Systolic pressure ≥150 millimeters of mercury (mmHg) and diastolic pressure ≥90 mmHg
  5. If proteinuria is ≥2+ in a qualitative test for urine protein, ≥1.0 grams for 24 hours is accumulated
  6. Complications or surgery (such as malabsorption syndrome, chronic diarrhea, or total gastrectomy) that could significantly influence the absorption of the investigational drug
  7. Have undergone major surgery within 4 weeks before enrollment
  8. Co-existing effusion requiring treatment
* Participants unable to take oral medication
* Participants scheduled for surgery during the projected course of the study
* Participants who test positive for human immunodeficiency virus (HIV antibody), or positive for hepatitis B surface (HBs antigen) or hepatitis C virus (HCV antibody)
* Participants who have taken lenvatinib before
* Participants who in the view of the principal investigator or sub-investigator are not able to comply with this protocol because of psychiatric or physical diseases including alcoholism or drug addiction
* Pregnant or nursing participants
* Participants who are participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve over the dosing interval on multiple dosing (AUC[0-τ]) | Day 1: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 2: pre-dose (24 hours after first administration). Day 8: pre-dose. Day 15: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 16: pre-dose (24 hours after administration on Day 15)
  Blood samples will be collected to determine the plasma lenvatinib concentration at the specified time points. AUC(0-τ) is defined as the area under the concentration-time profile from time zero to the end of the dosing interval at steady state. AUC represents the total drug exposure over a defined period of time.
Time at which the highest drug concentration occurs at steady-state (tss,max) | Day 1: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 2: pre-dose (24 hours after first administration). Day 8: pre-dose. Day 15: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 16: pre-dose (24 hours after administration on Day 15)
  Blood samples will be collected to determine the plasma lenvatinib concentration at the specified time points. tss,max is the time at which the maximum concentration of lenvatinib is observed in the plasma at steady state, which occurs when the rates of drug administration and drug elimination are equal.
Average steady-state concentration (Css,av) | Day 1: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 2: pre-dose (24 hours after first administration). Day 8: pre-dose. Day 15: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 16: pre-dose (24 hours after administration on Day 15)
  Blood samples will be collected to determine the plasma lenvatinib concentration at the specified time points. Css,av is the average concentration of lenvatinib in plasma at the time that a steady state has been achieved, which occurs when the rates of drug administration and drug elimination are equal.
Minimum observed concentration at steady-state (Css,min) | Day 1: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 2: pre-dose (24 hours after first administration). Day 8: pre-dose. Day 15: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 16: pre-dose (24 hours after administration on Day 15
  Blood samples will be collected to determine the plasma lenvatinib concentration at the specified time points. Css,min is the lowest concentration of lenvatinib in plasma at the time that a steady state has been achieved, which occurs when the rates of drug administration and drug elimination are equal.
Maximum observed concentration at steady-state (Css,max) | Day 1: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 2: pre-dose (24 hours after first administration). Day 8: pre-dose. Day 15: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 16: pre-dose (24 hours after administration on Day 15)
  Blood samples will be collected to determine the plasma lenvatinib concentration at the specified time points. Css,max is the highest concentration of lenvatinib in plasma at the time that a steady state has been achieved, which occurs when rates of drug administration and drug elimination are equal.
Area under the concentration-time curve from zero time to time of last quantifiable concentration (AUC[0-t]) | Day 1: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 2: pre-dose (24 hours after first administration). Day 8: pre-dose. Day 15: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 16: pre-dose (24 hours after administration on Day 15)
  Blood samples will be collected to determine the plasma lenvatinib concentration at various time points. AUC(0-t) is defined as the AUC from time "0" to the time of the last measurable concentration. AUC represents the total drug exposure over a defined period of time.
Time at which the highest drug concentration occurs (tmax) | Day 1: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 2: pre-dose (24 hours after first administration). Day 8: pre-dose. Day 15: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 16: pre-dose (24 hours after administration on Day 15)
  Blood samples will be collected to determine the plasma lenvatinib concentration at the specified time points. Tmax is the time at which the maximum concentration of lenvatinib is observed in plasma after a single dose of lenvatinib.
Maximum observed concentration (Cmax) | Day 1: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 2: pre-dose (24 hours after first administration). Day 8: pre-dose. Day 15: pre-dose; 1, 2, 4, and 8 hours post-dose. Day 16: pre-dose (24 hours after administration on Day 15)
  Blood samples will be collected to determine the plasma lenvatinib concentration at the specified time points. Cmax is the highest concentration of lenvatinib observed in plasma after a single dose of lenvatinib.

SECONDARY OUTCOMES:
Mean blood urea nitrogen (BUN) values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Blood samples will be collected to determine the amount of nitrogen in the blood.
Mean creatinine values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Blood chemistry tests will be performed to determine serum creatinine levels. Participants should be in a seated or supine position during blood collection.
Mean albumin values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Blood chemistry tests will be performed to determine serum albumin values. Participants should be in a seated or supine position during blood collection.
Mean cholesterol values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Blood chemistry tests will be performed to determine cholesterol levels. Participants should be in a seated or supine position during blood collection.
Mean lactate dehydrogenase values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Blood chemistry tests will be performed to determine serum lactate dehydrogenase levels. Participants should be in a seated or supine position during blood collection.
Mean total protein values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Blood chemistry tests will be performed to determine total protein levels. Participants should be in a seated or supine position during blood collection.
Mean C-reactive protein (CRP) values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Blood chemistry tests will be performed to determine CRP levels. Participants should be in a seated or supine position during blood collection.
Mean gamma-glutamyl transpeptidase (γ-GTP) values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Blood chemistry tests will be performed to determine γ-GTP levels. Participants should be in a seated or supine position during blood collection.
Mean total bilirubin values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Blood chemistry tests will be performed to determine total bilirubin levels. Participants should be in a seated or supine position during blood collection.
Mean alanine transaminase (ALT) values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  ALT is a transaminase enzyme and is commonly measured clinically as a biomarker for liver health. ALT will be summarized as the mean and standard deviation for all participants.
Mean aspartate transaminase (AST) values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  AST is a pyridoxal phosphate-dependent transaminase enzyme and is commonly measured clinically as a biomarker for liver health. AST will be summarized as the mean and standard deviation for all participants.
Mean alkaline phosphatase (ALP) values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  ALP is a hydrolase enzyme responsible for the dephosphorylation of molecules, including nucleotides, proteins, and alkaloids, and is commonly measured clinically as a biomarker for liver health. ALP will be summarized as the mean and standard deviation for all participants.
Mean body temperature | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Body temperature in degrees Celsius will be analyzed from the armpit of the participants. Body temperature will be summarized as the mean and standard deviation for all participants
Mean body weight | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Body weight of the participants will be measured in kilograms (kg). It will be summarized as the mean and standard deviation for all participants.
Mean heart rate | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Heart rate of the participants will be measured in beats per minute (bpm). It will be summarized as the mean and standard deviation for all participants.
Mean QT values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  The QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. QT values will be measured in milliseconds (msec) and will be summarized as the mean and standard deviation for all participants.
Mean QT corrected (QTc) values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  The QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. QTc values will be measured in milliseconds (msec) and it will be summarized as the mean and standard deviation for all participants.
Mean QTc corrected using Fridericia's method (QTcF) values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  The QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. QTcF values will be measured in msec and will be summarized as the mean and standard deviation for all participants.
Number of participants with abnormal, clinically significant physical examination findings | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Physical examinations will be performed to determine abnormal findings that meet the definition of an AE. Clinical significance will be determined by the Investigator.
Mean calcium values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Blood chemistry tests will be performed to determine calcium levels. Participants should be in a seated or supine position during blood collection.
Mean chloride values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Blood chemistry tests will be performed to determine chloride levels. Participants should be in a seated or supine position during blood collection.
Mean potassium values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Blood chemistry tests will be performed to determine potassium levels. Participants should be in a seated or supine position during blood collection.
Mean sodium values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Blood chemistry tests will be performed to determine sodium levels. Participants should be in a seated or supine position during blood collection.
Mean lymphocyte count | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Hematology tests will be performed to determine the lymphocyte count in blood. Participants should be in a seated or supine position during blood collection.
Mean neutrophil count | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Hematology tests will be performed to determine the neutrophil count in blood. Participants should be in a seated or supine position during blood collection.
Mean white blood cell (WBC) count | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Hematology tests will be performed to determine the WBC count in blood. Participants should be in a seated or supine position during blood collection.
Mean platelet count | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Hematology tests will be performed to determine the platelet count in blood. Participants should be in a seated or supine position during blood collection.
Mean hemoglobin values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Hematology tests will be performed to determine the hemoglobin levels in blood. Participants should be in a seated or supine position during blood collection.
Mean red blood cell (RBC) count | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Hematology tests will be performed to determine the RBC count in blood. Participants should be in a seated or supine position during blood collection.
Number of participants with any serious adverse event and any non-serious adverse event | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  An Adverse Event (AE) is any untoward medical occurrence in a clinical investigation participant administered with an investigational product. A serious adverse event (SAE) is any untoward medical occurrence that at any dose: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions; or is a congenital abnormality/birth defect.
Mean protein in urine values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Urine samples will be collected to determine the amount of protein in the urine.
Mean glucose in urine values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Urine samples will be collected to determine the amount of glucose in the urine.
Mean occult blood in urine values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Urine samples will be collected to determine the amount of microscopic blood in the urine.
Mean systolic blood pressure and diastolic blood pressure values | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Blood pressure will be measured after the participant has been sitting.
Mean pulse | until disease progression, development of unacceptable toxicity, participant requests to discontinue, or withdrawal of consent (up to Day 28)
  Pulse will be measured after the participant has been sitting.

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Information, Study Director — Eisai Inc.
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang

REFERENCES:
- [Derived] Liu D, Liu L, Shen L, Kubota T, Suzuki T, Ikezawa H, Shiba S, Bai Y. Pharmacokinetic study of lenvatinib in Chinese patients with solid tumors. Future Oncol. 2021 May;17(15):1855-1863. doi: 10.2217/fon-2020-0877. Epub 2021 Jan 21. PMID 33474967